CLINICAL TRIAL: NCT03538730
Title: Pain After Tonsillectomy Study
Acronym: PAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Melanie Noel, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB17-1794
Record Dates: First submitted 2018-04-02; First posted 2018-05-29 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: At 2-weeks post-surgery, parent-child dyads will participate in a lab visit during which time they will be randomized into an intervention or control group. Randomization will be conducted by an external statistician using a computer random number generator. Allocation concealment will be achieved using sequentially numbered, opaque, and sealed envelopes.
Who Masked: Participant, Outcomes Assessor
Masking Description: Group allocation will be revealed to one investigator at the outset of the lab visit. Other investigators and participants will remain masked until the end of the memory interview. Outcome assessors will remain masked for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control (No Intervention): Similar to previous narrative and memory interventions, parents in the control group will receive instructions from a researcher for 20 minutes on how to engage in child-directed play. Importantly, they will not talk about pain or the past surgery experience.
- Memory Reframing Intervention (Experimental): Parents in the intervention group will spend 20 minutes with a researcher and receive instructions about adaptive ways of reminiscing about the in-hospital and post-surgery periods.
  Interventions: Behavioral: Memory Reframing

INTERVENTIONS:
Behavioral: Memory Reframing — The intervention will draw from existing narrative-based interventions, past pain memory reframing interventions and findings from our recent data. Specifically, parents will be taught to reminisce with their children about the in-hospital and post-surgery periods by encouraging children to provide more explanations, using less utterances about pain, avoiding repetitions, emphasizing positive aspects of the child's surgery memory (e.g., when children used coping methods such as deep breathing, when they got a treat), and enhancing children's self-efficacy regarding their ability to cope with pain.
  Arms: Memory Reframing Intervention

SUMMARY:
Pain is a common experience in childhood. Healthy children can undergo up to 20 painful procedures by the age of 5. Moreover, millions of children undergo surgery (e.g., tonsillectomies) each year, which is commonly linked to pain and distress. Pain from, and fear of, medical experiences are not short lasting. Indeed, they can influence children long after the painful situation is over. Children's memories of pain after surgery can affect painful experiences in the future. Negative memories of pain (when children remember more pain than the actual level of pain experienced) are linked to higher pain and distress. As well, children who are more anxious and who experience greater pain are more likely to develop negatively biased pain memories, which then leads to greater fear and pain at subsequent pain experiences. It has been suggested that the ways in which parents and children talk about pain following painful events is important for how children remember the pain.

This study will be one of the first to look at whether a parent-led memory reframing intervention can reduce children's negative memories of surgery.

The study will include 100 children scheduled for a tonsillectomy and one of their parents. They will be recruited from the Alberta Children's Hospital. Parents will complete a survey 1-3 weeks before their child's surgery, and then the child's pain and anxiety will be monitored on the day of surgery and for 2 weeks after surgery. Two weeks after surgery, the parent and child will come to the hospital and be assigned to a control group or a memory reframing session. Six weeks after surgery, parents and children will complete a telephone interview.

DETAILED DESCRIPTION:
Background:

Pain is ubiquitous in childhood. Healthy children who are compliant with medical care undergo up to 20 painful procedures by the age of 5. Moreover, millions of children undergo surgery (e.g., tonsillectomies) each year, which is commonly linked to pain and distress. Pain from, and fear of, medical experiences can influence children long after the painful stimulus is removed. Children's memories of needle-related, experimental, post-surgical, and procedural pain are a powerful predictor of future pain experiences, even more so than the initial pain itself. Memory is susceptible to distortion. Negative biases in pain memories (i.e., recalled pain is higher than initial pain report) are associated with higher subsequent pain, distress, and worse medical compliance. Several factors have been implicated in the development of negatively biased pain memories in children. Higher child anxiety and pain are linked to negatively biased pain memories, which then leads to greater fear and pain at subsequent pain experiences. Parents and adolescents who think more catastrophically about child pain prior to surgery tend to develop more negatively biased pain memories months later. In fact, parents' catastrophic thinking about child pain was found to be the most important predictor of children's memory biases and subsequent pain trajectories.

Parental and child anxiety may lead to memory biases due to the ways in which parents and children discuss pain following painful events (e.g., by emphasizing threatening aspects of the experience). The investigators recently published a conceptual developmental framework in the journal PAIN outlining cognitive and social factors that may influence children's pain memory development. Of particular importance is early childhood (ages 4-7 years) when children are most prone to memory biases due to suggestibility effects. It is also during this time that parents are most influential in shaping children's cognitions, emotions, and behaviors. This model posits that the socio-linguistic context (e.g. parent-child narratives about pain) in which pain memories develop is most important in early childhood and sets the stage for future pain experiences.

There have been few studies examining memory reframing interventions in the context of children's recall of pain. In a recent systematic review, existing trials of memory reframing interventions were found to be efficacious in reducing negative memory biases. Parent-child reminiscing about past negative events plays a powerful role in how memories of those events are later retrieved and reframed. Parent-child narrative style also influences children's coping and psychological functioning. Young children of parents who are topic-extending and elaborative (e.g., who ask open-ended questions to pull for more detailed accounts of the past) and use emotional language, are more accurate and detailed in recalling their pasts, which is adaptive.

Recent data from the investigators' lab suggests that parents who reminisce with their children about surgery using a certain style (e.g., more elaborative, less topic-switching) and content (e.g., less content about pain, fear, medical procedures; more explanations) have children who later remember post-surgical pain in a more accurate or positively biased way. Parental reminiscing style and content have been effectively targeted in interventions to improve children's memory development. However, negatively biased memories of post-surgical pain, which can lead to persistent pain problems, have not been targeted, despite a need for interventions for this pediatric population. Moreover, existing memory reframing interventions did not employ parents. Parents are potentially the most powerful and accessible intervention agents, and the investigators' recent data provides strong evidence that the language parents use when reminiscing with children following surgery influences children's pain memory biases.

The aim of the proposed research study is to conduct a pilot study to examine the preliminary efficacy, feasibility, and acceptability of a brief parent-led memory reframing intervention following pediatric surgery to foster more adaptive (i.e., less negatively biased) pain memories. This study will be the first to develop and pilot test a brief, parent-led intervention aimed at changing the way children recall their pain after surgery. Given the vital role of pain memories in shaping future pain experiences and the need for interventions in the pediatric surgery context, this study has great potential to contribute an accessible and feasible post-surgical pediatric pain management intervention and foster more adaptive pain trajectories and medical experiences in childhood.

Study aims:

Primary Aim: To examine the preliminary efficacy, feasibility, and acceptability of a parent-led memory reframing intervention on children's post-surgical pain memories. Hypothesis 1: Children in the intervention group will go on to recall post-surgical pain in a more accurate or positively biased way as compared to the control group who will remember pain in a more negatively biased way. The intervention will be judged by parents to be feasible and acceptable.

Secondary Aim: To examine the influence of baseline individual child and parent characteristics on children's pain memories. Hypothesis 2: Children who are more anxious, less self-efficacious, have worse sleep quality, and whose parents are more anxious and catastrophize more about child pain prior to surgery will subsequently remember pain in a more negatively biased way.

Methods:

Sample:

One hundred children (50 intervention, 50 control) between the ages of 4-7 years and one of their parents will be recruited from the Ear Nose and Throat (ENT) Clinic at Alberta Children's Hospital.

Procedure:

Patients will be identified through surgery schedule lists. At entry into the clinic, a member of the ENT Clinic will provide potentially eligible patients with information about the study. Parents provide permission to be contacted by the research team. A few weeks before surgery, a member of the research team will conduct a recruitment phone call with all eligible patients' parents to discuss the study. After the recruitment phone call, online consent forms will be emailed to interested participants. Parents will provide consent for the child's participation; children, who are 7 years old or over or turn 7 during the course of participation in the study, will provide assent. One week before surgery, parents will complete measures of parent catastrophizing about child pain (PCS-P), child language (CCC2), and child sleep (SDSC). For descriptive purposes, parents will report on socio-demographics (e.g., child age, household income), preparation that they/their child received about the surgery, and family history of tonsillectomies and surgeries. On the day of surgery, measures of parental state anxiety (STAI-S) will be obtained as well as children's levels of pain intensity (FPS-R) and pain-related fear (CFS). A trained observer will objectively assess preoperative child anxiety during anesthesia induction (mYPAS).

As per standard clinical care: In Day Surgery, all patients will receive Tylenol 15 mg/kg orally pre-operatively, unless there is a specific contraindication. One parent may be present at anesthesia induction with their child. The child will receive an inhalational induction with sevoflurane, oxygen, and nitrous oxide. An intravenous will then be inserted, and the child will be maintained on either volatile anesthetic or total intravenous anesthetic (TIVA) for the procedure. During the procedure, all patients will receive dexamethasone 0.2 mg/kg IV, ondansetron 0.1 mg/kg IV, and morphine for analgesia. All of the ENT surgeons will use cautery to the tonsillar bed as their surgical technique for the procedure. The child will then be extubated deep or awake at the end of the procedure and transferred to the Post-Anesthesia Care Unit (PACU) to recover. Decision to bring a parent or caregiver into the PACU will be at the discretion of the PACU nurse and the anesthesiologist. Information regarding the surgical technique used and analgesic and anesthetic agents administered on the day of surgery will be collected via medical chart review.

A researcher will obtain ratings of child pain intensity and pain-related fear shortly following surgery. Parents will be given and instructed on how to administer these scales so that child-reports of pain can be captured at home. Proxy and self-reports of child average and worst pain intensity and pain-related fear will be assessed on days 1, 2, 3, 7 and 14 post-surgery. Proxy-reports of child sleep (SDSC) will be assessed on day 14 post-surgery. Parents will also report on the use of analgesics at home. At 2-weeks post-surgery, parents and children will come to the PI's research lab at the Alberta Children's Hospital during which time they will be randomized into an intervention or control group. Randomization will be conducted by an external statistician using a computer random number generator. Allocation concealment will be achieved using sequentially numbered, opaque, and sealed envelopes. Group allocation will be revealed by a researcher at the outset of the lab visit. During the lab visit, parents in both groups will talk to a researcher while another researcher plays with the child (e.g., coloring) in a separate room.

Control Group. Similar to previous narrative and memory interventions, parents in the control group will receive instructions from a researcher on how to engage in child-directed play. Importantly, they will not talk about pain or the past surgery experience. After this 20-minute period, parents in the control group will be instructed to reminisce with their children about the in-hospital and post-surgery periods as they normally would.

Intervention Group. Parents in the intervention group will receive instructions from a researcher about adaptive ways of reminiscing about the in-hospital and post-surgery periods. The intervention will draw from extant interventions that have taught parents to reminisce with their children about past negative events in more elaborative and emotion-rich ways (e.g., to use more open-ended questions, follow up on children's answers by providing new details about the event, talk more about emotions, and praise children's answers). Elements of past pain memory reframing interventions and findings from the investigators' recent data will also be included. Specifically, parents will be taught to reminisce with their children about the in-hospital and post-surgery periods by providing more explanations for events, using less utterances about pain, fear, and medical procedures, emphasizing positive aspects of the child's surgery memory, and enhancing children's self-efficacy regarding their ability to cope with pain. Researchers will also provide suggestions for specific questions and remarks to make while reminiscing. Parents and researchers will engage in brief role-plays to solidify the techniques, followed by researcher feedback. After this 20-minute period, parents in the intervention group will be instructed to reminisce with their children about the in-hospital and post-surgery periods using the intervention strategies.

After parents and children have finished reminiscing, parents in both groups will be asked to complete a short survey similar to the one completed at baseline. Three to four weeks after surgery, children in both groups will complete a telephone pain memory interview to assess children's recall of the in-hospital and post-surgery periods. Then, parents in the intervention group will complete a brief telephone interview to assess feasibility and acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo an elective outpatient tonsillectomy with or without adenoidectomy

Exclusion Criteria:

* Children receiving pre-medication with anxiolytics (Midazolam; administered to < 5% of youth),
* who have serious medical co-morbidities,
* and/or who have developmental disabilities or speech/language delays

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Memory | 3-4 weeks post-surgery
  Children will complete a pain memory interview via telephone where they will be asked to recall the in-hospital and post-surgery (i.e., while at home) time periods and complete the same pain intensity and pain-related fear scales based on their memories of those time periods. Biases in memory will be defined as the deviation in recalled and initial/experienced pain reports. Similar to our previous research, statistical models predicting pain memories will control for initial pain ratings that correspond to each memory question. Negatively biased pain memories will be defined as children who remember more pain and fear as compared to their initial pain reports. Positively biased pain memories will be defined as recalled pain that is less than initial pain reports. Accurate memories reflect no difference between recalled and experienced levels of pain.

SECONDARY OUTCOMES:
Child preoperative anxiety | Day of surgery
  The 27-item Modified Yale Preoperative Anxiety Scale (mYPAS) will be used by two trained observers to assess anxiety prior to and during anesthesia induction.
Child pain intensity | Day of surgery, days 1, 2, 3, 7, and 14 post-surgery, 3-4 weeks post-surgery
  We will capture sensory and affective aspects of pain and pain-related fear. Pain intensity will be assessed using a well-validated single-item faces pain scale (Faces Pain Scale-Revised; FPS-R), with anchors 'no pain' (0) and 'very much pain' (10).
Child pain-related fear | Day of surgery, days 1, 2, 3, 7, and 14 post-surgery, 3-4 weeks post-surgery
  We will capture sensory and affective aspects of pain and pain-related fear. Children's pain-related fear will be assessed using the Children's Fear Scale (CFS), with anchors 'not at all scared' (0) and 'most scared possible' (4).
Parent self-efficacy | 1 week pre-surgery, 2 weeks post-surgery
  Parents will rate their pain-related self-efficacy regarding their child's post-surgical pain using a single item 100-mm visual analogue scale (VAS). Parents will be asked to rate how confident they are that they could decrease their child's post-surgical pain, with anchors 'no confidence' (0) to 'complete confidence' (100).
Child sleep quality | 1 week pre-surgery, 2 weeks post-surgery
  The psychometrically-sound 26-item Sleep Disturbance Scale for Children (SDSC) will be used to assess parental report of children's sleep quality.
Child language and communication skills | 1 week pre-surgery
  The Children's Communications Checklist-2 (CCC-2) is a psychometrically-sound 70-item measure designed to assess communication skills in youth aged 4-16 years.
Parent anxiety | 1 week pre-surgery, day of surgery
  Parents will use the 40-item State-Trait Anxiety inventory (STAI) to assess their own state and trait anxiety.
Parent catastrophic thinking about child pain | 1 week pre-surgery, 2 weeks post-surgery
  The Pain Catastrophizing Scale-Parent Version (PCS-P) is a 13-item self-report measure that assesses catastrophic thoughts and feelings that parents may have when their child experiences pain.
Feasibility of intervention | 3-4 weeks post-surgery
  Feasibility will be assessed using study recruitment/enrollment statistics, completion of the study elements; and researchers' and parents' ratings of parents' motivation to learn, understanding of the intervention, and parent-child and parent-researcher rapport rated on 11-point Likert scales (0, 'not at all' to 10, 'very much').
Acceptability and satisfaction | 3-4 weeks post-surgery
  The parent-report 9-item Treatment Evaluation Inventory-Short Form (TEI-SF) will be used to assess parental acceptability and satisfaction with the intervention; however, items will be slightly modified to pertain to the memory reframing intervention.
Satisfaction of intervention | 3-4 weeks post-surgery
  Semi-structured telephone interviews will be conducted to assess treatment satisfaction (i.e., how parents felt about the intervention, if they liked it, if they think it worked, etc.) and elicit feedback.
Parent-child narratives | 2 weeks post-surgery
  Narratives will be video-recorded, transcribed, broken down into utterances, and coded by two independent coders using established coding schemes derived from the child development literature on children's narratives and memories. Coders have been trained and will be masked to treatment condition. The following aspects of narratives will be coded: Reminiscing style/level of elaboration (elaboration vs. repetition) and content (e.g., references to pain, anxiety/fear, medical procedures, emotions, explanations). Proportions of narrative utterance type over the entire number of utterances used will be calculated. Based on previous research, the primary narrative codes for the analyses will be parent reminiscing style (elaboration), and content related to pain, anxiety, medical procedures, and explanations.
Medical records review: Surgery technique | Day of surgery
  Through the medical records review, we will gather information about the surgery technique (Tonsillectomy, with or without adenoidectomy; additional procedures performed).
Medical records review: parental presence at induction | Day of surgery
  Through the medical records review, we will gather information about parental presence at induction (i.e., was a parent present? Yes/No).
Medical records review: anesthetic technique | Day of surgery
  Through the medical records review, we will gather information about the anesthetic technique (maintenance with volatile or TIVA), intraoperative opioid administration, awake or deep extubation.
Medical records review: duration of PACU stay | Day of surgery
  Through the medical records review, we will gather information about duration of PACU stay (in minutes).
Medical records review: parental presence in PACU | Day of surgery
  Through the medical records review, we will gather information about parental presence in PACU (i.e., was parent present in PACU? Yes/No).
Medical records review: analgesics in Day Surgery | Day of surgery
  Through the medical records review, we will gather information about analgesic administration in Day Surgery.
Medical records review: overnight stay | Day of surgery
  Through the medical records review, we will gather information about an overnight stay (i.e., did the child stay overnight after their surgery? Yes/No).
Analgesic consumption after discharge | Days 1, 2, 3, 7, and 14 post-surgery
  Analgesic administration (or absence thereof) will be recorded at home. The questions will include medicine type (including any specific remedies to reduce pain due to swallowing), dose, and number of times medicine was administered.
Socio-demographics | 1 week pre-surgery
  A brief socio-demographic form will be administered to assess: ethnic background, level of education, household income, and family composition.
Medical history | 1 week pre-surgery
  A brief medical history form will be administered to assess: family surgical and medical history, and surgery preparation and knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Noel, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavlova M, Lund T, Nania C, Kennedy M, Graham S, Noel M. Reframe the Pain: A Randomized Controlled Trial of a Parent-Led Memory-Reframing Intervention. J Pain. 2022 Feb;23(2):263-275. doi: 10.1016/j.jpain.2021.08.002. Epub 2021 Aug 21. PMID 34425247

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT03538730/Prot_SAP_000.pdf